CLINICAL TRIAL: NCT04381039
Title: The Effect of Customized Insoles on Biomechanics and Pain in Patients With Functional Flatfoot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201909067DINA
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Flexible Flatfoot
MeSH Terms: conditions — Flatfoot | interventions — Foot Orthoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- customized insole group (Experimental)
  Interventions: Device: Insole

INTERVENTIONS:
Device: Insole — 3D printing insole (Nylon), 3D printing insole (TPU), CNC machine insole (EVA), shoe only

SUMMARY:
The aim of present study is to compare the effects of 3D printing customized insoles using different thermoplastic materials on functional flatfoot patients' foot function and biomechanics

DETAILED DESCRIPTION:
Functional flatfoot is a common foot disease which induces pain and functional decline. Insoles can be used for intervention and correction, especially customized insoles which are made according to different foot types. There have been few studies using 3D printing for customized insoles for functional flatfoot. Besides, compared to traditional method and subtractive manufacturing, the effect of 3D printing customized insoles is still controversial and depends on technology, materials and design.The purpose of present study is to compare the effects of 3D printing customized insoles using different thermoplastic materials on functional flatfoot patients' foot function and biomechanics. Twelve patients with functional flatfoot (foot function index> 6) aged 20-65 years old will be recruited in this study. Participants plan to wear three kinds of customized insoles fabricated by 3D printing with Nylon and TPU or computer numerical control machine with EVA. F-Scan system and questionnaires will be used to record foot biomechanics and pain after wearing insoles immediately, and foot condition after three weeks. Statistical analysis will be adopted for repeated-measures analysis of variance （ANOVA） for all outcome measures and post-hoc test will be used to test the difference between groups.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 and 65 years old
* Appearance of decreased medial arch
* Foot posture index score between 6 to 12

Exclusion Criteria:

* History of injuries of the lower extremity within the past 6 months
* Experience of use of orthopedic insole within the past 6 months
* Acute disorders in the lower extremities and spine
* History of surgery on the lower extremities and lumbar spine within the past 6 months

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
F-scan system | after wearing insole (immediate effect)
  measure peak plantar pressure, contact area, peak force and center of pressure excursion index during walking and center of pressure velocity and center of pressure 95% ellipse area during one leg stance by F-scan system

SECONDARY OUTCOMES:
Visual analogue scale | after wearing insole (immediate effect)
  This scale is used to measure pain and wearing comfort during sitting, standing and walking. For pain measurement, the maximum value is 10, which means severe pain. The minimum value is 0, which means absence of pain. For comfort measurement, the maximum value is 10, which means most comfortable. The minimum value is 0, which means absence of comfort.
Foot function index | after wearing each insole for a week (at least 6 hours per day)
  Foot function index is used to measure foot condition. It contains 23 items, which are divided into three subscales: activity limitation, disability, and pain.
  The patient scores each question on a scale from 0 (no pain or difficulty) to 10 (worst pain imaginable or so difficult it requires help), that best describes their foot over the past week.
  Higher scores indicates worse pain. Both total and subcategory scores are calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Physical therapy center, national Taiwan university hosipital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No